CLINICAL TRIAL: NCT01656135
Title: Reference Group Trial for The ONE Study: A Unified Approach to Evaluating Cellular Immunotherapy in Solid Organ Transplantation
Brief Title: Reference Group Trial for The ONE Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Edward Geissler, Chief Investigator and EU Project Leader, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONErgt11; 260687 (Other Grant/Funding Number: EU FP7 Programme); 2011-004301-24 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: End-stage Renal Failure; Kidney Graft Rejection
Keywords: gold standard treatment; immune monitoring; acute rejection; graft rejection; living-donor; renal transplantation; kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection; Monitoring, Immunologic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reference Group (Other): Basiliximab (Simulect®):
  * Day 0: 20mg IV ≤2h prior to surgery
  * Day 4: 20mg IV
  Prednisolone:
  * Day 0: 500mg IV (250mg pre-op, 250mg intra-op)
  * Day 1: 125mg IV
  * Day 2 - 14: 20mg/day oral
  * Week 3 - 4: 15mg/day oral
  * Week 5 - 8: 10mg/day oral
  * Week 9 - 12: 5mg/day oral
  * Week 13 - 14: 2.5mg/day oral
  * Week 15 - Study End: Cessation
  Steroid tapering should not proceed if graft rejection has occurred or if renal dysfunction is observed.
  Mycophenolate Mofetil (MMF, or biologic equivalent):
  Treatment with MMF should commence one day prior to transplantation (on Day -1) and should continue indefinitely, with a dose reduction after two weeks:
  * Day -1 - 14: 2g/day oral
  * Day 15 - Study End 1.5g/day oral (750mg twice daily)
  Tacrolimus (or biologic equivalent):
  * Day -4 - 14: 3-12ng/ml
  * Week 3 - 12: 3-10ng/ml
  * Week 13 - 36: 3-8ng/ml
  * Week 37 - Study End: 3-6ng/ml
  Interventions: Other: Blood drawing for immune monitoring and questionnaires

INTERVENTIONS:
Other: Blood drawing for immune monitoring and questionnaires

SUMMARY:
To investigate the progression of the immunological response in living-donor kidney transplant recipients treated with a standard immunosuppressive regimen. Clinical, immunological, and health-economic data collected during this Reference Group Trial will be used to corroborate historical renal transplantation statistics and generate reference ranges for future clinical studies that will test immunoregulatory cell therapy as an adjunct immunosuppressive treatment in renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

Organ Donor:

A prospective donor is eligible for the research if all of the following inclusion criteria apply:

1. Eligible for live kidney donation
2. Aged at least 18 years
3. An ABO blood type compatible with the organ recipient
4. Willing and able to provide a blood sample for The ONE Study Subprojects
5. Willing to provide personal and medical/biological data for the trial
6. Signed and dated written informed consent.

In signing the donor information sheet/informed consent form (DIS/ICF), organ donors agree to provide a blood sample for the IM Subproject, and permit access to their medical records for the collection of specified demographic and medical/biological data for the trial.

Organ Recipient:

1. Chronic renal insufficiency necessitating kidney transplantation and approved to receive a primary kidney allograft from a living donor
2. Aged at least 18 years
3. Able to commence the immunosuppressive regimen at the protocol-specified time point
4. Willing and able to participate in The ONE Study subprojects
5. Signed and dated written informed consent.

Exclusion Criteria:

Organ Donor:

If a prospective donor fulfils any of the following criteria, then they are ineligible for the trial:

1. Genetically identical to the prospective organ recipient at the HLA loci
2. Exposure to any investigational agents at the time of kidney donation, or within 28 days prior to kidney donation
3. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
4. Subjects unable to freely give their informed consent (e.g. individuals under legal guardianship).

Organ Recipient:

1. Patient has previously received, or is scheduled to receive, any tissue or organ transplant other than the planned kidney graft
2. Known sensitivity to tacrolimus, mycophenolate, or corticosteroids
3. Genetically identical to the prospective organ donor at the HLA loci
4. PRA grade > 40% within 6 months prior to enrolment
5. Previous treatment with any desensitisation procedure (with or without IVIg)
6. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non-metastatic basal/squamous cell carcinoma of the skin)
7. Evidence of significant local or systemic infection
8. HIV-positive, EBV-negative or suffering chronic viral hepatitis
9. Significant liver disease, defined as persistently elevated AST and/or ALT levels >2 x ULN (Upper Limit of Normal range)
10. Malignant or pre-malignant haematological conditions
11. Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives
12. Any condition which, in the judgement of the Investigator, would place the subject at undue risk
13. Ongoing treatment with systemic immunosuppressive drugs at study entry
14. Participation in another clinical trial during the study or within 28 days prior to planned study entry
15. Female patients of child-bearing potential with a positive pregnancy test at enrolment
16. Female patients who are breast-feeding
17. All female patients of child-bearing potential UNLESS:

    1. The patient is willing to maintain a highly effective method of birth control for the duration of the study
    2. The career, lifestyle, or sexual orientation of the patient ensures that there is no risk of pregnancy for the duration of the study (at the discretion of the local Investigator)
18. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
19. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
20. Patients unable to freely give their informed consent (e.g. individuals under legal guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
biopsy-confirmed acute rejection incidence | 60 weeks

SECONDARY OUTCOMES:
time to first acute rejection episode | within 60 weeks
severity of acute rejection episodes | within 60 weeks
total immunosuppressive burden | 60 weeks
incidence of chronic graft dysfunction | 60 weeks
incidence of graft loss through rejection | 60 weeks
incidence of adverse drug reactions | 60 weeks
incidence of major infections | 60 weeks
incidence of neoplasia | 60 weeks
incidence of patients treated for subclinical acute rejection | 60 weeks

OTHER OUTCOMES:
Immune Monitoring (IM) assessment | 60 weeks
Health Economics (HEC) assessment | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward K. Geissler, Ph.D., Study Director — University of Regensburg
Locations (8):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- CHU de Nantes Hotel-Dieu, Nantes, France
- Germany (2):
  - Charite Campus Virchow-Klinikum, Berlin
  - University Hospital Regensburg, Regensburg
- Ospedale San Raffaele, Milan, Italy
- United Kingdom (2):
  - Guy's Hospital in affiliation with King's College London, London
  - Churchill Hospital in affiliation with the University of Oxford, Oxford

REFERENCES:
- [Derived] Sly LM, McKay DM. Macrophage immunotherapy: overcoming impediments to realize promise. Trends Immunol. 2022 Dec;43(12):959-968. doi: 10.1016/j.it.2022.10.002. Epub 2022 Oct 29. PMID 36441083
- [Derived] Moreau A, Kervella D, Bouchet-Delbos L, Braudeau C, Saiagh S, Guerif P, Limou S, Moreau A, Bercegeay S, Streitz M, Sawitzki B, James B, Harden PN, Game D, Tang Q, Markmann JF, Roberts ISD, Geissler EK, Dreno B, Josien R, Cuturi MC, Blancho G; DIVAT consortium. A Phase I/IIa study of autologous tolerogenic dendritic cells immunotherapy in kidney transplant recipients. Kidney Int. 2023 Mar;103(3):627-637. doi: 10.1016/j.kint.2022.08.037. Epub 2022 Oct 26. PMID 36306921
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407
- See also: The ONE Study — http://www.onestudy.org